CLINICAL TRIAL: NCT06514404
Title: Comparative Study of Empathy and Anxiety in the Different Academic Years, at the Beginning of Academic Year and Exam Period and the Relationship of These Variables With Personality at the University of León and Madrid in the Degree of Nursing, Physiotherapy and Podiatry.
Brief Title: Comparative Study of Empathy and Anxiety in the Different Academic Years, at the Beginning of Academic Year and Exam Period in Healthy Students.
Status: Not yet recruiting | Type: Observational
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Profesor, Universidad Complutense de Madrid
Other Study IDs: C.I. 23/792-E
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Health Education; Health Promotion; Health Behavior
Keywords: health students; anxiety; empahty; assessment personality; Health behavior
MeSH Terms: conditions — Health Education; Health Behavior; Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — Observational study of the effects on anxiety and empathy of personality the situation of start academic year in health sciences

SUMMARY:
Students from different health science degrees will carry out a study on the variables of empathy, anxiety and personality profile.

DETAILED DESCRIPTION:
Students from different health science degrees will carry out a study on the variables of empathy, anxiety and personality profile by means of validated questionnaires in order to compare them between different Spanish regions and in different courses to be able to see their evolution and characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are studying a health grade.
* Subjects that wish to participate in the study.

Exclusion Criteria:

* Students who do not wish to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — we will compare the students by sex
Study Population: Health science students are the target population of this study and the aim is to obtain data on their state and trait anxiety as well as its relationship with personality at the beginning of the academic year.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Empathy Quotent | Through study completion, an average of 1 week
  It consists of 60 items, 40 measuring empathy and 20 control measures. Scores range from 0 to 80. It measures cognitive and affective empathy in adults. Equalizer allows classification into four categories, which facilitates comparison between groups. The cut-off for each level is: from 0 to 32 scores: low empathy (average scores in Asperger Syndrome is 20), from 33 to 52 scores: average empathy (average in men 42, average in women 47), from 53 to 63 scores: above average, from 64 to 80 scores: high empathy
State anxiety | Through study completion, an average of 1 week
  The response scale is Likert-type with 4 alternatives (in the Spanish adaptation from 0 to 3). There are 20 items for evaluation. Thus, the range of responses goes from 0 to 60, with a higher level of anxiety corresponding to a higher score.
Anxiety as a trait | Through study completion, an average of 1 week
  The response scale is Likert-type with 4 alternatives (in the Spanish adaptation from 0 to 3). Trait anxiety has 20 items for its evaluation. Thus, the range of responses goes from 0 to 60, with a higher level of anxiety corresponding to a higher score.
Abbreviated personality questionnaire | Through study completion, an average of 1 week
  The EPQR-A is an abbreviated form of the Eysenck Personality Questionnaire. It is a 24-item self-report measure that leverages three personality scales (extraversion, neuroticism and psychoticism) and a lie validity scale. Each scale is assessed by 6 questions that participants rate on a binary frequency scale scored 1 or 0.

IPD SHARING:
Plan to Share IPD: No